CLINICAL TRIAL: NCT05373771
Title: Sickle Cell Improvement: Enhancing Care in the Emergency Department
Acronym: SCIENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Pediatric Emergency Care Applied Research Network (Network); Nemours Children's Health System (Other)
Responsible Party: Principal Investigator, David Brousseau, Professor, Chair, Nemours Children's Health System
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 00114249
Record Dates: First submitted 2022-05-05; First posted 2022-05-13 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Sickle Cell Crisis
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-intervention (Active Comparator)
  Interventions: Other: Care pathway
- Delayed intervention (No Intervention)

INTERVENTIONS:
Other: Care pathway — Implementation of care pathway as part of hybrid type 2 implementation effectiveness study
  Arms: Post-intervention

SUMMARY:
Sickle cell disease (SCD) is an inherited blood disorder affecting approximately 36,000 children in the United States, approximately 90% of whom are Black. The disease is characterized by recurrent, severe pain crises which result in high rates of emergency department visits and hospitalizations, and decreased quality of life. The National Heart, Lung and Blood Institute, as well as the American Society of Hematology, have endorsed pain management guidelines regarding the timeliness of care for children presenting with these acute pain crises. These evidence-based guidelines are infrequently followed, resulting in increased pain and hospitalizations. In additional to other barriers to following the guideline, structural racism has been proposed as a significant contributor and the New England Journal of Medicine recently called for the institution of SCD-specific pain management protocols to combat structural racism and reduce time to opioid administration. The investigators' long-term goal is to improve the care and health outcomes of children with acute painful vaso-occlusive crisis treated in the emergency department. The overall aim of the investigators is to test a care pathway using multifaceted implementation strategies to increase guideline adherent care for children in the emergency department with acute painful vaso-occlusive crisis.

ELIGIBILITY:
Inclusion Criteria:

* ED visit for uncomplicated pain crisis
* Sickle cell disease
* Receipt of at least one opioid

Exclusion Criteria:

* Acute chest syndrome
* Fever > 38.5 in the ED
* priapism
* sickle cell trait

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5328 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Timeliness of receipt of opioids | A maximum of about 6 hours as all opioids received during the ED stay will be captured
  The percent of patients who receive first dose of opioids within 60 minutes of arrival and subsequent doses within 30 minutes of previous dose

SECONDARY OUTCOMES:
Median time to opioids | A maximum of about 6 hours as all opioids received during the ED stay will be captured
  Median time from arrival to first opioid and then subsequent opioids
Percent of children hospitalized | A maximum of about 6 hours as that is the typical maximum time to disposition for patients
  Disposition of hospitalization or discharge home

CONTACTS AND LOCATIONS:
Overall Officials: David Brousseau, MD, MS, Principal Investigator — Nemours Children's Health
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Outcome data gathered through central data Registry. It is a limited dataset. A public use dataset will be made available after the study consistent with NIH guidelines.